CLINICAL TRIAL: NCT04984278
Title: A Randomized, Double-blind, Placebo-controlled, 2-way Crossover Trial to Evaluate the Effect of Nabiximols Oromucosal Spray on Clinical Measures of Spasticity in Patients With Multiple Sclerosis
Brief Title: Evaluation of the Effect of Nabiximols Oromucosal Spray on Clinical Measures of Spasticity in Participants With Multiple Sclerosis
Acronym: RELEASE MSS5
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated based on a business decision by the Sponsor.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GWSP20105; 2020-003271-18 (EudraCT Number)
Record Dates: First submitted 2021-07-14; First posted 2021-07-30 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Spasticity With Multiple Sclerosis
Keywords: multiple sclerosis; MS; spasticity; velocity-dependent muscle tone; nabiximols
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nabiximols (Experimental): Nabiximols is a complex botanical medicine formulated from extracts of the cannabis plant that contains the principal cannabinoids delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD) and also contains minor constituents, including other cannabinoid and non-cannabinoid plant components, such as terpenes, sterols, and triglycerides. Study dependent: Each spray delivers 100 microliters (μL) of nabiximols. A pre-determined number of sprays, but no less than 4 sprays, of nabiximols will be self-administered by participants as an oromucosal spray, under supervision of trial staff during 2 study visits to the trial site after they temporarily discontinued treatment with prescribed nabiximols (Sativex) as part of their regular medication.
  Interventions: Drug: Nabiximols
- Placebo (Placebo Comparator): Placebo to match nabiximols is presented as an oromucosal spray containing the excipients ethanol and propylene glycol (50% v/v) with colorings and flavored with peppermint oil (0.05% v/v). Each spray delivers 100 μL containing no active ingredients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nabiximols — oromucosal spray
  Other Names: GW-1000-02; Sativex
  Arms: Nabiximols
Drug: Placebo — oromucosal spray
  Arms: Placebo

SUMMARY:
This study will be conducted to evaluate the effect of multiple doses of nabiximols compared with placebo on a clinical measure of velocity-dependent muscle tone in the lower limbs (Lower Limb Muscle Tone-6 [LLMT-6]) in participants with multiple sclerosis (MS). LLMT-6 is defined as the average of the 6 individual Modified Ashworth Scale (MAS)-transformed scores of knee flexors, knee extensors, and plantar flexors on both sides of the body.

DETAILED DESCRIPTION:
Each period of this multicenter, randomized, double-blind, placebo-controlled, 2-treatment, 2-period, crossover trial includes a 7-day Baseline period, a 3-week treatment period (comprising a 2-week titration phase and a 1-week maintenance phase).

Eligible participants will enter the 7-day baseline period of each treatment period. During baseline, participants will maintain their optimized oral MS antispasticity medication regimen and record their 11-point Numerical Rating Scale (NRS) spasticity score and spasm count using an electronic daily diary. On Day 1, eligible participants will be randomized to 1 of 2 treatment sequences, each composed of 2 treatment periods, with administration of multiple doses of nabiximols or placebo in a 1:1 ratio.

Participants will be advised to titrate the investigational medicinal product (IMP), beginning with 1 spray/day, to an optimized dose or to a maximum of 12 sprays/day over the first 14 days of treatment. Participants should continue at the same dose level achieved at the end of the titration phase ±1 spray divided into a morning dose and an evening dose for the remainder of the treatment period.

Lower limb muscle tone, health-related quality of life, safety, tolerability, and pharmacokinetics will be evaluated during the treatment period.

Participants who complete the trial will participate for a total of approximately 11 weeks (77 days), including the 7-day baseline period.

ELIGIBILITY:
Inclusion Criteria:

Screening (Visit 1)

* Willing and able to give informed consent for participation in the trial
* Willing and able (in the investigator's opinion) to comply with all trial requirements
* Has had a diagnosis with any disease subtype of multiple sclerosis (MS), by revised 2017 McDonald criteria, for at least 12 months prior to Visit 1 (Screening) and is expected to remain stable for the duration of the trial
* Has an Modified Ashworth Scale (MAS) untransformed score of at least 2 in 2 or more of 6 muscle groups (right knee flexors, left knee flexors, right knee extensors, left knee extensors, right plantar flexors, or left plantar flexors) at Visit 1 (Screening)
* If currently receiving approved anti-spasticity therapy, it must be with a stable dosing regimen for at least 30 days prior to Visit 1 (Screening). The participant must be willing to maintain the same antispasticity medication and not plan to initiate a new course of physiotherapy for the duration of the trial.
* If currently receiving an approved MS disease-modifying therapy, it must be at a stable dose for at least 3 months prior to Visit 1 (Screening) and be expected to remain stable for the duration of the trial.
* If currently receiving dalfampridine or fampridine, it must be at a stable dose for at least 3 months prior to Visit 1 (Screening) and is expected to remain stable for the duration of the trial.

Additional Inclusion Criteria at Randomization (Visit 2)

- Completed at least 5 of 7 days of their electronic diary reporting during the 7 days immediately preceding Visit 2 (Day 1)

Exclusion Criteria:

* Has taken nabiximols, cannabis, or a cannabis-derived product for medicinal or recreational purposes in the 30 days prior to Visit 1 (Screening) or unable to abstain for the duration of the study
* Did not tolerate or did not respond adequately to treatment with nabiximols or another cannabis-based medication if exposed at any time before the 30-day period prior to Visit 1 (Screening)
* Any concomitant disease or disorder that has spasticity-like symptoms or that may influence the participant's level of spasticity
* Medical history suggests that relapse/remission is likely to occur during the trial, which, in the opinion of the investigator, is expected to influence the participant's spasticity
* Has had a relapse of MS within the 60 days prior to Visit 1 (Screening)
* Currently using botulinum toxin injection for the relief of spasticity (within 6 months of Visit 1 [Screening]) or is unwilling to abstain for the duration of the trial
* Currently taking antipsychotic medication
* Currently taking benzodiazepines unless doses and dosing regimen have been stable for at least 30 days prior to Visit 1 (Screening)
* Clinically suspected to have a contracture in one of the muscle groups of the lower limbs, preventing assessment with the MAS
* Has any known or suspected hypersensitivity to cannabinoids or any of the excipients of the investigational medicinal product (IMP)
* Male and fertile (i.e., after puberty unless permanently sterile by bilateral orchiectomy) unless willing to ensure that he uses male contraception (condom or vasectomy) or remains sexually abstinent during the trial and for 3 months thereafter
* Female and of childbearing potential (i.e., following menarche and until becoming postmenopausal for ≥ 12 consecutive months unless permanently sterile by hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) unless willing to ensure that she uses a highly effective method of birth control (e.g., intrauterine device/hormone-releasing system, bilateral tubal occlusion, vasectomized partner, or sexual abstinence) during the trial and for 3 months thereafter. Participants using combined hormonal methods or a progestogen-only pill or injection or implant should use an additional barrier method such as a male condom or diaphragm during the trial and for 3 months thereafter.
* Female and pregnant (positive pregnancy test at Visit 1 [Screening] or Visit 2 [Day 1]), lactating, or planning pregnancy during the course of the trial or within 3 months thereafter.
* Has received an IMP within the 30 days prior to Visit 1 (Screening)
* Has any other clinically significant disease or disorder (including seizure disorder) that, in the opinion of the investigator, may put the participant, other participants, or site staff at risk because of participation in the trial, influence the interpretation of trial results, or may affect the participant's ability to take part in the trial
* Has any abnormalities identified following a physical examination, clinical laboratory, serology, or other applicable screening procedures that, in the opinion of the investigator, would jeopardize the safety of the participant or the conduct of the study if he or she took part in the trial
* Has any history of suicidal behavior in the 5 years prior to Visit 1 (Screening) or a score of 3, 4, or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the month prior to Visit 1 (Screening)
* Has any known or suspected history of alcohol or substance abuse (including opiate abuse) or dependence within 1 year prior to Visit 1 (Screening)
* Currently using an illicit drug or current nonprescribed use of any prescription drug
* Has a history of psychiatric or neurologic disorder that, in the opinion of the investigator, may interfere with trial participation, data interpretation, or conduct of trial procedures
* Has a history of severe psychiatric disorder that may be exacerbated by the use of a cannabinoid-containing product
* Has any planned clinical interventions or intends to change any or all medications that may have an effect on spasticity or MS during the trial
* Currently taking drugs that are solely metabolized by UGT1A9 and UGT2B7
* Currently taking strong CYP3A4 inducers (e.g., rifampicin, carbamazepine, phenytoin, phenobarbital, St. John's Wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (6):
  - Mountain View Clinical Research, Denver, Colorado
  - Collier Neurologic Specialists, Naples, Florida
  - University of South Florida, Tampa, Florida
  - Consultants in Neurology - Northbrook, Chicago, Illinois
  - Premier Neurology Research, PC, Greer, South Carolina
  - Neurology Clinic-Cordova, Cordova, Tennessee
- Czechia (3):
  - NeuropsychiatrieHK, Choceň
  - NeuropsychiatrieHK, Hradec Králové
  - Krajská Zdravotní - Nemocnice Teplice, Teplice
- Poland (12):
  - Niepubliczny Zakład Opieki Zdrowotnej NEURO - KARD, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne Neuromed - Ośrodek Badań Klinicznych, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Małopolskie Centrum Kliniczne, Krakow, Lesser Poland Voivodeship
  - Instytut Zdrowia dr Boczarska-Jedynak, Oświęcim, Lesser Poland Voivodeship
  - Indywidualna Praktyka Lekarska Dr Hab Konrad Rejdak, Lublin, Lublin Voivodeship
  - Centrum Medyczne Pratia - Warszawa, Warsaw, Masovian Voivodeship
  - Szpital Wolski im dr. Anny Gostyńskiej Samodzielny Publiczny Zakład Opieki Zdrowotnej, Warsaw, Masovian Voivodeship
  - MA-LEK A.M. Maciejowscy S.C. Centrum Terapii SM, Katowice, Silesian Voivodeship
  - DENDRYT Centrum Medyczne, Katowice, Silesian Voivodeship
  - Neuro-Medic Janusz Zbrojkiewicz, Katowice, Silesian Voivodeship
  - Wielospecjalistyczne Centrum Medyczne Ibismed, Zabrze, Silesian Voivodeship
  - RESMEDICA Poradnia Neurologiczna, Kielce, Świętokrzyskie Voivodeship
- Spain (4):
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Institut Hospital del Mar d'Investigacions Mèdiques, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Vithas Nisa Sevilla, Seville
- United Kingdom (5):
  - Panthera Biopartners - North London, North London, England
  - ReCognition Health - Plymouth, Plymouth, England
  - Panthera Biopartners - Preston, Preston, England
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, England
  - NHS Highland, Inverness, Scotland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 31 participants who met all inclusion criteria and no exclusion criteria were randomized to treatment at 7 clinic centers in Poland, Czech Republic, Spain, and United Kingdom.
Pre-assignment Details: After signing the ICF, participants with spasticity associated with MS participated in a Screening Period of up to 28 days; changes in the dosing regimen of the participants' current MS antispasticity medications, if any, were not made during this period.
Groups:
- Nabiximols First, Then Placebo: Participants who were randomized to receive GW-1000-02 (nabiximols) self-administered as an oromucosal spray for 21 days (starting on Day 1; Treatment Period 1), followed by at least a 7-day wash out period, and then received matching placebo treatment for 21 days (starting at Day 31; Treatment Period 2). For each treatment period, participants titrate the investigational medicinal product (IMP), beginning with 1 spray/day, to an optimized dose or to a maximum of 12 sprays/day over the first 14 days of treatment and then continue at the same dose level ±1 spray, divided into a morning dose and an evening dose for the remainder of the treatment period.
- Placebo First, Then Nabiximols: Participants who were randomized to receive matching placebo self-administered as an oromucosal spray for 21 days (starting on Day 1; Treatment Period 1), followed by at least a 7-day wash out period, and then received GW-1000-02 (nabiximols) treatment for 21 days (starting at Day 31; Treatment Period 2). For each treatment period, participants titrate the investigational medicinal product (IMP), beginning with 1 spray/day, to an optimized dose or to a maximum of 12 sprays/day over the first 14 days of treatment and then continue at the same dose level ±1 spray, divided into a morning dose and an evening dose for the remainder of the treatment period.
Period: Period 1
Arm/Group | Nabiximols First, Then Placebo | Placebo First, Then Nabiximols
Started | 16 | 15
Completed | 15 | 14
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 0 | 1
Period: Period 2
Arm/Group | Nabiximols First, Then Placebo | Placebo First, Then Nabiximols
Started | 15 | 14
Completed | 14 | 13
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed in the Full Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nabiximols First, Then Placebo | Placebo First, Then Nabiximols | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (10.3) | 48.8 (7.4) | 51.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lower Limb Muscle Tone-6 (LLMT-6)
Description: LLMT-6 is defined as the average of the 6 individual Modified Ashworth Scale (MAS) transformed scores of knee flexors, knee extensors, and plantar flexors on both sides of the body. Transformed MAS ranges from 0 (no increase in muscle tone) to 5 (affected part rigid in flexion or extension). The combined (treatment period 1 and treatment period 2) least square mean change from baseline in LLMT-6 score is being reported. Negative values indicate an improvement in muscle tone.
Time Frame: Baseline (predose Day 1 of Treatment Period 1) up to Day 51 (end of treatment of Treatment Period 2)
Population: LLMT-6 was assessed in the Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Nabiximols: A 21-day treatment period with nabiximols self-administered as an oromucosal spray (without regard to treatment period).
- Placebo: A 21-day treatment period with placebo self-administered as an oromucosal spray (without regard to treatment period).
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | -0.32 (0.072) | -0.04 (0.075)
Statistical Analysis 1: Comparison: Nabiximols vs Placebo; Test type: Superiority; p = 0.0048, Mixed Models Analysis; Combined least mean square difference = -0.29, 95% CI 2-sided [-0.48 to -0.10], Standard Error of Mean 0.092

2. Secondary Outcome: Change From Baseline in Lower Limb Muscle Tone-4 (LLMT-4)
Description: LLMT-4 is defined as the average of the 4 individual MAS transformed scores of knee flexors and knee extensors on both sides of the body. Transformed MAS ranges from 0 (no increase in muscle tone) to 5 (affected part rigid in flexion or extension). The combined (treatment period 1 and treatment period 2) least square mean change from baseline in LLMT-4 score is being reported. Negative values indicate an improvement in muscle tone.
Time Frame: Baseline (predose Day 1 of Treatment Period 1) up to Day 51 (end of treatment of Treatment Period 2)
Population: LLMT-4 was assessed in the Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | -0.34 (0.079) | -0.09 (0.082)

3. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is an adverse event that started, or worsened in severity or seriousness, following the first dose of the investigational medicinal product.
Time Frame: Baseline (predose Day 1 of Treatment Period 1) up to Day 51 (end of treatment of Treatment Period 2)
Population: TEAEs were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 30 | 30
Participants | 19 | 6

4. Secondary Outcome: Change From Baseline in Blood Pressure
Time Frame: Baseline (predose Day 1 of Treatment Period 1) up to Day 51 (end of treatment of Treatment Period 2)
Population: Vital signs were assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 29 | 27
mmHg
  Systolic blood pressure | -2.5 (11.27) | -4.4 (8.26)
  Diastolic blood pressure | -1.9 (7.74) | -2.8 (7.66)

5. Secondary Outcome: Change From Baseline in Heart Rate
Time Frame: Baseline (predose Day 1 of Treatment Period 1) up to Day 51 (end of treatment of Treatment Period 2)
Population: Vital signs were assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 29 | 27
beats/minute | 0.9 (8.97) | -0.1 (9.13)

6. Secondary Outcome: Change From Baseline in Clinical Laboratory Test Values
Time Frame: Baseline (predose Day 1 of Treatment Period 1) up to Day 51 (end of treatment of Treatment Period 2)
Population: Clinical laboratory tests were assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 27 | 25
10^9 cells per liter
  Leukocytes | 0 (1.68) | -0.07 (1.94)
  Neutrophils: number analyzed (Participants) | 15 | 12
  Neutrophils | 0.071 (0.94) | -0.399 (0.53)
  Basophils | -0.01 (0.07) | 0 (0.07)
  Eosinophils | 0.04 (0.22) | 0.04 (0.19)
  Lymphocytes | -0.041 (0.48) | 0.033 (0.48)
  Monocytes | 0.01 (0.22) | 0.03 (0.20)
  Platelets | 2.4 (23.20) | 4.6 (25.91)

7. Secondary Outcome: Change From Baseline in Erythrocytes
Time Frame: Baseline (predose Day 1 of Treatment Period 1) up to Day 51 (end of treatment of Treatment Period 2)
Population: Clinical laboratory tests were assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 27 | 27
10^12 cells per liter | -0.138 (0.20) | -0.090 (0.19)

8. Secondary Outcome: Change From Baseline in Hemoglobin
Time Frame: Baseline (predose Day 1 of Treatment Period 1) up to Day 51 (end of treatment of Treatment Period 2)
Population: Clinical laboratory tests were assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 27 | 25
g/dL | -0.34 (0.62) | -0.21 (0.53)

9. Secondary Outcome: Change From Baseline in Hematocrit Ratio
Description: Hematocrit was measured in whole blood samples. The ratio of packed cells to total volume was assessed. Normal ratio ranges from 0.350-0.470 female and 0.400-0.540 male (normal ranges per our central lab), 0.37 (or 37%) to 0.52 (or 52%) in adults. Lower hematocrit ratios indicate worse clinical outcome.
Time Frame: Baseline (predose Day 1 of Treatment Period 1) up to Day 51 (end of treatment of Treatment Period 2)
Population: Clinical laboratory tests were assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: ratio of packed cells to total volume
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 27 | 25
ratio of packed cells to total volume | -0.012 (0.0191) | -0.009 (0.0191)

10. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Volume
Time Frame: Baseline (predose Day 1 of Treatment Period 1) up to Day 51 (end of treatment of Treatment Period 2)
Population: Clinical laboratory tests were assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 27 | 25
fL | -0.12 (2.08) | -0.38 (1.89)

11. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Hemoglobin
Time Frame: Baseline (predose Day 1 of Treatment Period 1) up to Day 51 (end of treatment of Treatment Period 2)
Population: Clinical laboratory tests were assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 27 | 25
pg | 0.1 (0.64) | 0.1 (0.57)

12. Secondary Outcome: Change From Baseline in Electrocardiogram Parameters
Time Frame: Baseline (predose Day 1 of Treatment Period 1) up to Day 51 (end of treatment of Treatment Period 2)
Population: Electrocardiogram parameters were assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 29 | 27
msec
  PR duration | -3.1 (27.35) | 0.5 (26.78)
  QRS duration | 2.0 (6.10) | 1.7 (5.54)
  QT interval | 5.4 (15.35) | 4.0 (17.79)
  QTcB interval | -0.8 (16.04) | 4.9 (15.20)
  QTcF interval | 2.5 (12.60) | 5.2 (13.84)

13. Secondary Outcome: Change From Baseline in Electrocardiogram Pulse Rate
Time Frame: Baseline (predose Day 1 of Treatment Period 1) up to Day 51 (end of treatment of Treatment Period 2)
Population: Vital signs were assessed in the Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 29 | 27
beats/minute | -2.0 (9.42) | -0.1 (7.78)

14. Secondary Outcome: Number of Participants With Suicidal Ideation or Behavior Based on The Columbia Suicide Severity Rating Scale (CSSRS)
Description: The C-SSRS is a short questionnaire that is used to assess suicidal ideation (5 questions) and behavior (5 questions) since last patient visit. The questionnaire is completed by participants answering yes or no to each question.
Time Frame: Baseline, Day 15, and Day 21
Population: Suicidal ideation or behavior was assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 30 | 30
Participants
  Baseline, Suicidal ideation | 0 | 0
  Baseline, Suicidal ideation, Wish to be dead | 0 | 0
  Baseline, Suicidal ideation, Non-specific active suicidal thoughts | 0 | 0
  Baseline, Suicidal ideation, Active with any methods (not planned) without intent to act | 0 | 0
  Baseline, Suicidal ideation, Active with some intent to act, without specific plan | 0 | 0
  Baseline, Suicidal ideation, Active with specific plan and intent | 0 | 0
  Baseline, Suicidal behavior | 0 | 0
  Baseline, Suicidal behavior, Preparatory acts or behavior | 0 | 0
  Baseline, Suicidal behavior, Aborted attempt | 0 | 0
  Baseline, Suicidal behavior, Interrupted attempt | 0 | 0
  Baseline, Suicidal behavior, Actual attempt (non-fatal) | 0 | 0
  Baseline, Suicidal behavior, Completed suicide | 0 | 0
  Baseline, Suicidal ideation or behavior | 0 | 0
  Baseline, Self-injurious behavior without suicidal intent | 0 | 0
  Day 15, Suicidal ideation | 0 | 1
  Day 15, Suicidal ideation, Wish to be dead | 0 | 0
  Day 15, Suicidal ideation, Non-specific active suicidal thoughts | 0 | 0
  Day 15, Suicidal ideation, Active with any methods (not planned) without intent to act | 0 | 1
  Day 15, Suicidal ideation, Active with some intent to act, without specific plan | 0 | 1
  Day 15, Suicidal ideation, Active with specific plan and intent | 0 | 0
  Day 15, Suicidal behavior | 0 | 0
  Day 15, Suicidal behavior, Preparatory acts or behavior | 0 | 0
  Day 15, Suicidal behavior, Aborted attempt | 0 | 0
  Day 15, Suicidal behavior, Interrupted attempt | 0 | 0
  Day 15, Suicidal behavior, Actual attempt (non-fatal) | 0 | 0
  Day 15, Suicidal behavior, Completed suicide | 0 | 0
  Day 15, Suicidal ideation or behavior | 0 | 0
  Day 15, Self-injurious behavior without suicidal intent | 0 | 0
  Day 21, Suicidal ideation | 0 | 0
  Day 21, Suicidal ideation, Wish to be dead | 0 | 0
  Day 21, Suicidal ideation, Non-specific active suicidal thoughts | 0 | 0
  Day 21, Suicidal ideation, Active with any methods (not planned) without intent to act | 0 | 0
  Day 21, Suicidal ideation, Active with some intent to act, without specific plan | 0 | 0
  Day 21, Suicidal ideation, Active with specific plan and intent | 0 | 0
  Day 21, Suicidal behavior | 0 | 0
  Day 21, Suicidal behavior, Preparatory acts or behavior | 0 | 0
  Day 21, Suicidal behavior, Aborted attempt | 0 | 0
  Day 21, Suicidal behavior, Interrupted attempt | 0 | 0
  Day 21, Suicidal behavior, Actual attempt (non-fatal) | 0 | 0
  Day 21, Suicidal behavior, Completed suicide | 0 | 0
  Day 21, Suicidal ideation or behavior | 0 | 0
  Day 21, Self-injurious behavior without suicidal intent | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event (TEAE) data were collected from baseline (predose Day 1 of Treatment Period 1) up to Day 51 (end of treatment of Treatment Period 2).
Description: A TEAE is an adverse event that started, or worsened in severity or seriousness, following the first dose of the investigational medicinal product.
Arm/Group | Nabiximols | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 6/30 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nabiximols (N=30) | Placebo (N=30)
Vertigo (Ear and labyrinth disorders) | 2 | 0
Fatigue (General disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT04984278/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT04984278/SAP_001.pdf